CLINICAL TRIAL: NCT03393403
Title: Comparison of the Effect of Intravenous Continuous Dexmedetomidine Infusion and Dexmedetomidine as a Local Anesthetic Adjuvant in Subcostal Transverse Abdominis Plane Block in Patients Undergoing Gastric Cancer Surgery
Brief Title: Comparison of the Effect of Intravenous and Perineural Dexmedetomidine in Gastric Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, KMUHIRB-F(II)-20170001, Physician, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20170001
Record Dates: First submitted 2017-12-27; First posted 2018-01-08 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Gastric Cancer; Pain, Postoperative
Keywords: Subcostal transversus abdominis plane block
MeSH Terms: conditions — Stomach Neoplasms; Pain, Postoperative | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine_iv group (Experimental): Dexmedetomidine 0.5mcg/kg (diluted in normal saline) intravenously infusion for 30min
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine_adj group (Experimental): Dexmedetomidine 0.5mcg/kg (adding to local anesthetic) perineural single bolus for subcostal TAP block 0.9% sodium chloride 0.125ml/kg intravenously infusion for 30min
  Interventions: Drug: Dexmedetomidine; Drug: 0.9% Sodium-chloride
- Control group (Active Comparator): 0.9% sodium chloride 0.125ml/kg intravenously infusion for 30min No dexmedetomidine use
  Interventions: Drug: 0.9% Sodium-chloride

INTERVENTIONS:
Drug: Dexmedetomidine — 0.5mcg/kg intravenous(IV)continuous infusion for 30 minutes, or 0.5mcg/kg adding to local anesthetic for subcostal TAP block
  Other Names: Precedex
  Arms: Dexmedetomidine_adj group; Dexmedetomidine_iv group
Drug: 0.9% Sodium-chloride — 0.125ml/kg intravenously infusion in Dexmedetomidine_adj group and control group
  Arms: Control group; Dexmedetomidine_adj group

SUMMARY:
Using random case assignment to investigate the analgesic and sedative effect of intravenous dexmedetomidine and dexmedetomidine as a local anesthetic adjuvant in ultrasound-guided subcostal TAP block in gastric cancer patient undergoing gastrectomy or partial gastrectomy.

DETAILED DESCRIPTION:
The process of the experiment (brief describe) The participant patients will be randomly allocated into three groups: the intravenous dexmedetomidine group (Dex_iv group), dexmedetomidine adding to local anesthetic as an adjuvant for subcostal TAP block (Dex_adj group), and Control group. All patients receive gastrectomy or partial gastrectomy in general anesthesia as standard. Thirty minutes before the end of surgery, the patients in Dex_iv group receive 0.5mcg/kg dexmedetomidine infusion for 30 minutes, while the patients in Dex_adj group and control group receive 0.125ml/kg 0.9% normal saline IV infusion for 30 minutes. All patients have ultrasound-guided TAP block single injection after the end of surgery and before the tracheal tube extubation. The block agents in Dex_adj group is 40 ml of 0.375% ropivacaine with 0.5mcg/kg dexmedetomidine, while in Dex_iv group and control group are only 40ml of 0.375% ropivacaine. The IV PCA pump will be set up before patients awaken in the post-anesthesia care unit. All patients are assessed for the signs of emergence agitation with Riker sedation-agitation scale in the post-anesthesia care unit. The numerical rating scale (NRS) for pain intensity assessment, the opioid consumption via IV PCA pump, and the patients satisfaction will be documented for postoperative 3 days for the impact evaluation of dexmedetomidine in postoperative analgesia in patients undergoing gastric cancer surgery with subcostal TAP block.

ELIGIBILITY:
Inclusion Criteria:

* gastric cancer patients undergoing gastrectomy or partial gastrectomy, who receive ultrasound-guided subcostal TAP block and PCA for postoperative analgesia

Exclusion Criteria:

* surgery involved other visceral organ (eg. combined splenectomy or partial hepatectomy), patients with histories of adverse drug reaction to dexmedetomidine, bradycardia (baseline heart rate <60 beats/min), any type of atrioventricular block in electrocardiogram (EKG), heart failure, significant renal or hepatic impairment, severe bronchopulmonary disease, any coagulant disorder, and pregnant or breast-feeding woman.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-12-23 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
analgesic effect - pain intensity | postoperative 3 days
  postoperative acute pain intensity (numerical rating scale, NRS, 0-10)

SECONDARY OUTCOMES:
sedative effect | postoperative 2 hours
  emergence agitation in post-anesthesia care unit (Riker sedation-agitation scale, 1-7)
analgesic effect - opioid consumption | postoperative 3 days
  Fentanyl consumption(mcg) via patient-control analgesia (PCA) pump

CONTACTS AND LOCATIONS:
Overall Officials: Miao-Pei Su, M.D., Principal Investigator — Physician
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No